CLINICAL TRIAL: NCT05641454
Title: The Effect of a Peat and Apple Extract on Muscle ATP and Exercise Performance
Acronym: APEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: VDF FutureCeuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 516252
Record Dates: First submitted 2022-11-01; First posted 2022-12-07 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Caffeine and Endurance Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ElevATP supplement (Experimental)
  Interventions: Dietary Supplement: ElevATP supplement
- Maltodextrin placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ElevATP supplement — ElevATP supplement containing apple and ancient peat extract
  Arms: ElevATP supplement
Dietary Supplement: Placebo — Maltodextrin placebo
  Arms: Maltodextrin placebo

SUMMARY:
A study to test the hypothesis that a combined peat and apple extract will increase blood and muscle ATP, which will increase cycling performance

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40
* Healthy
* Recreationally active (i.e. Participants will be deemed as too trained if they are defined as participating in structured resistance exercise 3 or more times per week for >6 months or participating in structured endurance exercise for >6h per week for >6 months. Participants will be defined as too sedentary if they do not exceed the governments guidelines of 150 / 75 min per week of light / heavy exercise.)

Exclusion Criteria:

* Allergy to Lidocaine
* Any diagnosed metabolic health condition
* Pregnant
* Non-habitual caffeine intake
* Smoker
* Diagnosed Cardiovascular disease
* Beta-Blockers
* Recent history of musculoskeletal injury

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Muscle ATP concentration | 4 hours
  Concentration of ATP in skeletal muscle tissue (mmol/kg dry weight)

SECONDARY OUTCOMES:
Total work performed during exercise | 2 hours
  Work performed during glycogen depleting exercise on a cycle ergometer (J)
Blood ATP concentration | 4 hours
  Concentration of ATP in blood (mmol/L)
Substrate oxidation | 1 hour
  Substrate oxidation over 1 h steady state cycle (g/min)
Blood glucose concentration | 4 hours
  Concentration of glucose in blood (mmol/L)
Blood lactate concentration | 4 hours
  Concentration of lactate in blood (mmol/L)
Muscle glycogen | 4 hours
  Muscle glycogen concentration in skeletal muscle tissue (mmol/kg dry weight)
Muscle ADP concentration | 4 hours (mmol/kg dry weight)
  Concentration of muscle metabolites
Muscle ATP concentration | 4 hours (mmol/kg dry weight)
  Concentration of muscle metabolites
Muscle creatine concentration | 4 hours (mmol/kg dry weight)
  Concentration of muscle metabolites
Muscle phosphocreatine concentration | 4 hours (mmol/kg dry weight)
  Concentration of muscle metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No